CLINICAL TRIAL: NCT00697385
Title: Open Label Continuation Study for the Use of Cyclokapron for Treatment and Management of Women With Bleeding Disorders
Brief Title: The Use of Cyclokapron for Treatment and Management of Women With Bleeding Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary M. Gooley Hemophilia Center (Other)
Responsible Party: Peter A. kouides, M.D., Mary M. Gooley Hemophilia Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 758-A-03-1
Record Dates: First submitted 2008-06-10; First posted 2008-06-13 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: vonWillebrand Disease; Hemophilia; Platelet Coagulation Disorders
MeSH Terms: conditions — Hemophilia A | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TA (Experimental): on treatment
  Interventions: Drug: Cyclokapron

INTERVENTIONS:
Drug: Cyclokapron — (2) 500mg tablets taken by mouth every 6-8 hours
  Other Names: tranexamic Acid

SUMMARY:
The high percentage of failure using available non-surgical options to treat menorrhagia in women with bleeding disorders shows a continuing need for innovative treatments. This has led to development of this protocol in order to make available tranexamic acid as a potentially effective menorrhagia therapy option in women with an underlying bleeding disorder. We anticipate that Tranexamic Acid may be a beneficial choice for controlling menorrhagia in bleeding disorder patients.

DETAILED DESCRIPTION:
Women with heavy periods and with a diagnosed bleeding disorders are prescribed cyclokapron pills to be taken during their periods. Their periods are assessed at 3 and 6 months by filling out a pictorial blood assessment chart. If the drug appears to be working with no adverse effects the patients can continue to take the medication as long as it is available with follow up with the investigator every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* all menstruating women regardless of age
* Women with heavy periods as measured by pictorial blood assessment chart
* Women diagnosed with a bleeding disorder

Exclusion Criteria:

* Acquired defective color vision
* Factor VIII, Factor IX, FactorXI levels >250%
* An inherited thrombophilic defect detected because of a positive family or personal history of thrombosis
* Current use of oral contraceptives

Ages: 8 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2003-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Reduced pictorial blood assessment chart scores from baseline | 3 and 6 months after start of medication

SECONDARY OUTCOMES:
increased hematocrit | 3 and 6 months from start of medication

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Kouides, MD, Principal Investigator — Mary M. Gooley Hemophilia Center
Locations (1):
- Mary M. Gooley Hemophilia Center, Rochester, New York, United States